CLINICAL TRIAL: NCT01987895
Title: A Multi-center, Randomized, Double-blind Study to Compare the Efficacy and Safety of Cadazolid Versus Vancomycin in Subjects With Clostridium Difficile-associated Diarrhea (CDAD)
Brief Title: Efficacy and Safety of Cadazolid Versus Vancomycin in Subjects With Clostridium Difficile - Associated Diarrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-061A301
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Clostridium Difficile Infection
Keywords: Post-antibiotic diarrhea; Clostridium difficile infection
MeSH Terms: conditions — Clostridium Infections | interventions — cadazolid; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cadazolid (Experimental): Subjects receive oral cadazolid 250 mg twice daily (bid) and oral vancomycin-matching placebo 4 times per day (qid) for 10 days
  Interventions: Drug: Cadazolid; Drug: Vancomycin-matching placebo
- Vancomycin (Active Comparator): Subjects receive oral vancomycin 125 mg qid and oral cadazolid-matching placebo bid for 10 days
  Interventions: Drug: Vancomycin; Drug: Cadazolid-matching placebo

INTERVENTIONS:
Drug: Cadazolid — Cadazolid 250 mg as oral suspension twice daily.
  Other Names: ACT-179811
  Arms: Cadazolid
Drug: Vancomycin — Vancomycin 125 mg as oral capsules 4 times daily.
  Other Names: Vancocin
  Arms: Vancomycin
Drug: Cadazolid-matching placebo — Placebo matching cadazolid and administered orally twice daily
  Arms: Vancomycin
Drug: Vancomycin-matching placebo — Placebo capsules matching vancomycin and administered orally 4 times per day
  Arms: Cadazolid

SUMMARY:
This clinical study is conducted to assess the efficacy of cadazolid compared to vancomycin in subjects with Clostridium difficile-associated diarrhea (CDAD).

DETAILED DESCRIPTION:
Subjects selected to participate in the study are treated either with cadazolid or vancomycin for 10 days. At the end of treatment, clinical cure is assessed; subjects are then followed-up to assess any disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent.
* Male or female ≥ 18 years of age. Females of childbearing potential must agree to use an adequate and reliable method of contraception.
* Subject with a diagnosis of mild-moderate or severe CDAD (first occurrence or first recurrence within 3 months) with: Diarrhea: a change in bowel habits with > 3 liquid or unformed bowel movements (UBM) within 24 hours prior to randomization, AND Positive C. difficile toxin test on a stool sample produced within 72 hours prior to randomization.

Exclusion Criteria:

* More than one previous episode of CDAD in the 3-month period prior to randomization.
* Evidence of life-threatening or fulminant CDAD.
* Likelihood of death within 72 hours from any cause.
* History of inflammatory colitides, chronic abdominal pain, or chronic diarrhea.
* Antimicrobial treatment active against CDAD administered for > 24 hours except for metronidazole treatment failures (MTF)
* Known hypersensitivity or contraindication to study drugs, oxazolidinones, or quinolones.
* Unable or unwilling to comply with all protocol requirements.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2017-02-26 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Claire Marrast, MD, Study Director — Actelion

REFERENCES:
- [Derived] Gerding DN, Cornely OA, Grill S, Kracker H, Marrast AC, Nord CE, Talbot GH, Buitrago M, Gheorghe Diaconescu I, Murta de Oliveira C, Preotescu L, Pullman J, Louie TJ, Wilcox MH. Cadazolid for the treatment of Clostridium difficile infection: results of two double-blind, placebo-controlled, non-inferiority, randomised phase 3 trials. Lancet Infect Dis. 2019 Mar;19(3):265-274. doi: 10.1016/S1473-3099(18)30614-5. Epub 2019 Jan 29. PMID 30709665
- [Derived] Kleinman L, Talbot GH, Hunsche E, Schuler R, Nord CE. The CDI-DaySyms: Content Development of a New Patient-Reported Outcome Questionnaire for Symptoms of Clostridium difficile Infection. Value Health. 2018 Apr;21(4):441-448. doi: 10.1016/j.jval.2017.08.3017. Epub 2017 Nov 7. PMID 29680101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 904 patients at 70 sites in 12 countries were screened, among whom 632 were enrolled in the IMPACT 1 trial at 64 sites located in North & South America, Europe and Australia.
Groups:
- Cadazolid: Subjects with Clostridium difficile-associated diarrhea (CDAD) received oral cadazolid 250 mg twice daily (bid) and oral vancomycin-matching placebo 4 times a day (qid) for 10 days. Subjects were followed up for 30 days after the last dose of cadazolid. Subjects who had a first recurrence of CDAD during the follow-up period were offered to enter a re-treatment extension period with cadazolid (10 day of cadazolid + 30-day follow up)
- Vancomycin: Subjects with CDAD received oral vancomycin 125 mg qid and oral cadazolid-matching placebo bid for 10 days. Subjects were followed up for 30 day after the last dose of vancomycin. Subjects who had a first recurrence of CDAD during the follow-up period were offered to enter a re-treatment extension period with cadazolid (10 day of cadazolid + 30-day follow up)
Period: Overall Study
Arm/Group | Cadazolid | Vancomycin
Started | 306 | 326
Completed (Include subjects who completed the main study + subjects who completed the re-treatment extension.) | 276 | 296
Not Completed | 30 | 30
Not completed — Withdrawal by Subject | 12 | 7
Not completed — Physician Decision | 8 | 10
Not completed — Death | 7 | 7
Not completed — Lost to Follow-up | 3 | 5
Not completed — randomized before giving IC | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline characteristics were defined using the modified intent-to-treat analysis set (mITT) including all randomized subjects who have received at least one dose of the study drug and had a confirmed diagnosis of CDAD
Groups:
- Total: Total of all reporting groups
Arm/Group | Cadazolid | Vancomycin | Total
Number analyzed (Participants) | 302 | 318 | 620
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 180 | 203 | 383
  65-74 years | 73 | 70 | 143
  75 years and older | 49 | 45 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 195 | 378
  Male | 119 | 123 | 242
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 9 | 12
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 288 | 299 | 587
  Other | 2 | 4 | 6
  Missing | 6 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101 | 108 | 209
  Canada | 83 | 88 | 171
  Europe | 111 | 117 | 228
  Other | 7 | 5 | 12
CDAD episode type strata [Count of Participants; unit: Participants] — CDAD episode type strata was defined as baseline stratification factor 'First occurrence' or 'First recurrence' of CDAD as recorded in the Interactive voice recognition system (IVRS) at the time of subject randomization. Number of subjects with first recurrence or first occurrence at randomization was assessed for each treatment group.
  Participants
    First occurrence | 238 | 253 | 491
    First recurrence | 64 | 65 | 129
Initial strain of Clostridium difficile [Count of Participants; unit: Participants] — The strain of C. difficile at baseline was identified in the last stool sample collected up to treatment start date and with available C. difficile culture. Identification was done by polymerase chain reaction (PCR). The strains were categorized as hypervirulent strains (PCR ribotype 027, 078 or 244) or non-hypervirulent (other PCR ribotypes). The number of subjects with hypervirulent, non-hypervirulent strains at baseline was assessed for each treatment group. If PCR ribotype at baseline was not available, the subjects were classified as "unable to determine".
  Participants
    Hypervirulent strains | 58 | 82 | 140
    Non-hypervirulent strains | 226 | 215 | 441
    Unable to determine | 18 | 21 | 39
CDAD severity at baseline [Count of Participants; unit: Participants] — CDAD at baseline was considered as severe if the following criteria were met: maximum body temperature > 38.5 C, white blood cell counts > 15.0 x 10*9/L and rise in baseline serum creatinine > 50% compared to the level before CDAD diagnosis. Otherwise, it was considered as mild-moderate. The number of subjects with severe and mild-moderate CDAD at baseline was assessed for each treatment group. If any of the measurements required for derivation of severity was missing, the subjects were classified as "unable to determine".
  Participants
    Mild-Moderate | 227 | 243 | 470
    Severe | 59 | 51 | 110
    Unable to determine | 16 | 24 | 40

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate (CCR) in the Modified Intent-to-treat Population
Description: Clinical Cure (CC) is defined as: • Resolution of Diarrhea (≤ 3 unformed bowel movement per day for at least 2 consecutive days) on study treatment and maintained for 2 days after end-of-treatment (EOT), AND • No additional antimicrobial treatment active against Clostridium difficile-associated diarrhea (CDAD) or fecal microbiota transplant between first dose of study drug and 2 days after EOT.
  CCR is the percentage of subjects with Clinical Cure. Analyses are performed on two analysis sets. Results on the modified intent-to-treat set (mITT) are reported below.
Time Frame: Up to Day 12 on average (end-of-treatment + 2 days)
Population: All subjects who received at least one dose of study drug and had a confirmed diagnosis of CDAD.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 302 | 318
Percentage of participants | 83.8 [79.2 to 87.5] | 85.2 [80.9 to 88.7]
Statistical Analysis 1: Comparison: Cadazolid vs Vancomycin; Test type: Non-Inferiority — Non-inferiority of CCR for cadazolid versus vancomycin is demonstrated if the lower limit of the 95% confidence interval (CI) is above -10%; Difference between 2 proportions = -1.4, 95% CI 2-sided [-7.2 to 4.3] — CI for the difference between two proportions are estimated using the Wilson's score method
Statistical Analysis 2: Comparison: Cadazolid vs Vancomycin; Sensitivity analysis with imputation for a single day with missing UBM data between one day before end-of-treatment (EOT) and 2 days after EOT; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference between 2 proportions = -2.4, 95% CI 2-sided [-8.1 to 3.2] — CI for the difference between two proportions are estimated using the Wilson's score method

2. Primary Outcome: Clinical Cure Rate (CCR) in the Per-protocol Population
Description: Clinical Cure (CC) is defined as: • Resolution of Diarrhea (≤ 3 unformed bowel movement per day for at least 2 consecutive days) on study treatment and maintained for 2 days after end-of-treatment (EOT), AND • No additional antimicrobial treatment active against Clostridium difficile-associated diarrhea (CDAD) or fecal microbiota transplant between first dose of study drug and 2 days after EOT. CCR is the percentage of subjects with Clinical Cure. Analyses are performed on two analysis sets. Results on the per-protocol set (PPS) are reported below.
Time Frame: Up to Day 12 on average (end-of-treatment + 2 days)
Population: All subjects who received at least one dose of study drug and had a confirmed diagnosis of CDAD and without protocol deviations that might affect the evaluation of the effect of the study drug on the primary variable.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 282 | 288
Percentage of participants | 87.6 [83.2 to 90.9] | 91.7 [87.9 to 94.3]
Statistical Analysis 1: Comparison: Cadazolid vs Vancomycin; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference between 2 proportions = -4.1, 95% CI 2-sided [-9.2 to 1.0] — CI for the difference between two proportions are estimated using the Wilson' score method

3. Secondary Outcome: Sustained Cure Rate (SCR) in the Modified Intent-to-treat Population
Description: Sustained Cure is defined for each subject having Clinical Cure and no recurrence. SCR is the percentage of subjects with Sustained Cure. The main analysis is performed on the modified intent-to-treat set (mITT).
Time Frame: Between Day 38 and Day 42 on average (end-of-treatment + 28-32 days)
Population: All subjects who received at least one dose of study drug and had a confirmed diagnosis of CDAD.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 302 | 318
Percentage of participants | 65.6 [60.0 to 70.7] | 62.3 [56.8 to 67.4]
Statistical Analysis 1: Comparison: Cadazolid vs Vancomycin; Test type: Superiority — Superiority of cadazolid versus vancomycin is demonstrated if the lower limit of the 95% confidence interval (CI) is above zero; Difference between 2 proportions = 3.3, 95% CI 2-sided [-4.3 to 10.8] — CI for the difference between two proportions are estimated using the Wilson's score method

4. Secondary Outcome: Kaplan-Meier Estimates for Resolution of Diarrhea
Description: Resolution of Diarrhea (ROD) is defined as no more than 3 unformed bowel movements per day for at least two consecutive days for subjects on study treatment.
  The Kaplan-Meier estimates (KM estimates) for having an event (ROD) are reported for each time point.
Time Frame: Up to Day 10
Population: The analyses were performed on the modified intention-to-treat population: all subjects who received at least one dose of study drug and had a confirmed diagnosis of CDAD
Measure: Number (95% Confidence Interval); unit: KM estimate (%)
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 302 | 318
KM estimate (%)
  Day 1 | 46.7 [41.2 to 52.5] | 45.9 [40.6 to 51.6]
  Day 2 | 62.6 [57.2 to 68.0] | 60.7 [55.4 to 66.1]
  Day 3 | 69.9 [64.6 to 74.9] | 71.1 [66.0 to 76.0]
  Day 4 | 72.8 [67.7 to 77.7] | 77.7 [73.0 to 82.1]
  Day 5 | 77.8 [73.0 to 82.3] | 80.2 [75.6 to 84.4]
  Day 6 | 81.1 [76.5 to 85.3] | 81.8 [77.3 to 85.8]
  Day 7 | 82.5 [78.0 to 86.5] | 84.6 [80.4 to 88.3]
  Day 8 | 83.4 [79.0 to 87.4] | 85.2 [81.1 to 88.9]
  Day 9 | 83.8 [79.4 to 87.7] | 85.2 [81.1 to 88.9]
  Day 10 | 83.8 [79.4 to 87.7] | 85.2 [81.1 to 88.9]
Statistical Analysis 1: Comparison: Cadazolid vs Vancomycin; Test type: Superiority; p = 0.6016, Log Rank — two-sided p-value (alpha 5%) based on log-rank test stratified by first occurrence / first recurrence and geographical region; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.80 to 1.14]

5. Secondary Outcome: Change From Baseline to Day 3 in Clostridium Difficile Infection (CDI) Daily Symptoms Patient-Reported Outcome (CDI-DaySyms PRO) Domain Scores
Description: CDI-DaySyms PRO is a questionnaire assessing 10 symptoms relevant to subjects with CDAD and grouped into 3 domains: Diarrhea symptoms, Abdominal symptoms and Systemic/Other. The subjects rate the severity of each item as None, Mild, Moderate, Severe or Very severe, converted to numeric scores from 0 to 4, respectively. The daily domain score is calculated as the mean of the non-missing responses for that domain on that day. A negative value for change from baseline corresponds to an improvement in domain score. The three domains are evaluated in a hierarchical manner, starting with Diarrhea Symptoms, then Abdominal Symptoms, and finally Systemic/Other Symptoms. The least squares means (LSM) are computed on the scores.
Time Frame: Day 1 (baseline) and Day 3
Population: All subjects from the modified intent-to-treat population, excluding those who participated in the validation sub-study. No imputation of missing scores is performed prior to deriving response status. Subjects with missing values at baseline or at Day 3 are considered to be non-responders.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 246 | 260
Score on a scale
  Diarrhea symptoms | -1.233 [-1.37 to -1.09] | -1.235 [-1.37 to -1.10]
  Abdominal symptoms | -0.623 [-0.74 to -0.51] | -0.710 [-0.82 to -0.60]
  Other symptoms | -0.639 [-0.74 to -0.54] | -0.689 [-0.79 to -0.59]
Statistical Analysis 1: Comparison: Cadazolid vs Vancomycin; Comparison of the diarrhea domain scores; Test type: Superiority; p = 0.9814, ANOVA — Two-sided 5% alpha level was used; ANOVA for repeated measurements was fitted using all values from Day 1 (baseline) to Day 12; Least Square Mean difference = 0.002, 95% CI 2-sided [-0.20 to 0.20] — The Least Square Means of the treatments differences for the changes from baseline at Day 3 were obtained using estimate statements
Statistical Analysis 2: Comparison: Cadazolid vs Vancomycin; Comparison of the abdominal symptoms domain scores; Test type: Superiority; p = 0.2879, ANOVA — Two-sided 5% alpha level was used; ANOVA for repeated measurements was fitted using all values from Day 1 (baseline) to Day 12; Least Square Mean difference = 0.087, 95% CI 2-sided [-0.07 to 0.25] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Cadazolid vs Vancomycin; Comparison of the systemic / other symptoms domain scores; Test type: Superiority; p = 0.4880, ANOVA — Two-sided 5% alpha level was used; ANOVA for repeated measurements was fitted using all values from Day 1 (baseline) to Day 12; Least Square Mean difference = 0.050, 95% CI 2-sided [-0.09 to 0.19] — [estimate comment as in outcome 5, analysis 1]

6. Other Pre Specified Outcome: Investigator's Assessment of Clinical Response (ICR) Rate at Visit 4 in the Modified Intent-to-treat Population
Description: ICR rate (%) is the percentage of subjects with clinical response assessed as cured according to the investigator's own judgement. Subjects with missing assessment are considered as not cured for the analysis. ICR rate is used as a supportive measure of the primary efficacy endpoint (CCR). Analyses are performed on two analysis sets. Results on the modified intent-to-treat set (mITT) are reported below.
Time Frame: Up to Day 12 on average (up to end-of-treatment + 2 to 4 days)
Population: All subjects who received at least one dose of study drug and had a confirmed diagnosis of CDAD.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 302 | 318
Percentage of participants | 89.7 [85.8 to 92.7] | 91.5 [87.9 to 94.1]
Statistical Analysis 1: Comparison: Cadazolid vs Vancomycin; Exploratory analysis; Test type: Other; Difference between 2 proportions = -1.8, 95% CI 2-sided [-6.5 to 2.9] — CI for the difference between two proportions are estimated using the Wilson's score method

7. Other Pre Specified Outcome: Investigator's Assessment of Clinical Response (ICR) Rate at Visit 4 in the Per-protocol Population
Description: ICR rate (%) is the percentage of subjects with clinical response assessed as cured according to the investigator's own judgement. ICR rate (%) is the percentage of subjects with ICR assessed as cured. Subjects with missing assessment are considered as not cured for the analysis. ICR rate is used as a supportive measure of the primary efficacy endpoint (CCR). Analyses are performed on two analysis sets. Results on the per-protocol set (PPS) are reported below.
Time Frame: Up to Day 12 on average (up to end-of-treatment + 2 to 4 days)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 282 | 288
Percentage of participants | 92.2 [88.5 to 94.8] | 94.1 [90.8 to 96.3]
Statistical Analysis 1: Comparison: Cadazolid vs Vancomycin; Exploratory analysis; Test type: Other; Difference between 2 proportions = -1.9, 95% CI 2-sided [-6.2 to 2.3] — CI for the difference between two proportions are estimated using the Wilson's score method

8. Other Pre Specified Outcome: Investigator's Assessment of Sustained Response Rate (ISR Rate) at Visit 5
Description: ISR rate (%) is the percentage of subjects assessed as Sustained Cure at Visit 5, according to the investigator's own judgement. Sustained Cure is defined for each subject having Clinical Cure and no recurrence. Subjects with missing assessment are considered as having 'Not Sustained Cure' for the analysis.
  ISR rate is used as a supportive measure of the secondary efficacy endpoint (SCR). Analyses are performed on the modified intent-to-treat set (mITT).
Time Frame: Between Day 38 and Day 42 on average (end-of-treatment + 28 to 32 days)
Population: All subjects who received at least one dose of study drug and had a confirmed diagnosis of CDAD.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 302 | 318
Percentage of participants | 73.8 [68.6 to 78.5] | 70.1 [64.9 to 74.9]
Statistical Analysis 1: Comparison: Cadazolid vs Vancomycin; Exploratory analysis; Test type: Other; Difference between 2 proportions = 3.7, 95% CI 2-sided [-3.4 to 10.7] — CI for the difference between two proportions are estimated using the Wilson's score method

9. Other Pre Specified Outcome: Sustained Cure Rate (SCR) in the Per-protocol Population
Description: Sustained Cure is defined for each subject having Clinical Cure and no recurrence. SCR is the percentage of subjects with Sustained Cure. The analyses performed on the modified intent-to- treat set (mITT) are repeated on the per-protocol set (PPS) for sensitivity.
Time Frame: Between Day 38 and Day 42 on average (end-of-treatment + 28-32 days)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 282 | 288
Percentage of participants | 68.8 [63.2 to 73.9] | 67.7 [62.1 to 72.8]
Statistical Analysis 1: Comparison: Cadazolid vs Vancomycin; Test type: Other — Sensitivity analysis; Difference between 2 proportions = 1.1, 95% CI 2-sided [-6.5 to 8.7] — CI for the difference between two proportions are estimated using the Wilson's score method

10. Other Pre Specified Outcome: Recurrence Rate
Description: Recurrence is defined as the occurrence of a new episode of diarrhea (> 3 unformed bowel movements on any day between end-of-treatment + 3 days and end-of-treatment + 30 days ) Recurrence rates is the percentage of subjects assessed as having a recurrence out of subjects with Clinical Cure.
Time Frame: Between Day 13 and Day 40 on average (from end-of-treatment + 3 days and end-of-treatment + 30 days)
Population: Subjects from the modified intent-to-treat analysis set with clinical cure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cadazolid | Vancomycin
Number analyzed (Participants) | 253 | 271
percentage of participants | 15 [11.1 to 19.9] | 21.4 [16.9 to 26.7]

ADVERSE EVENTS:
Time Frame: Serious and frequent adverse events are reported from study treatment initiation up to Day 17 on average (i.e., 7 days after end-of-treatment or study withdrawal) and all-cause mortality up to Day 40 on average (i.e. 28 to 32 days after end-of-treatment or study withdrawal)
Groups:
- Cadazolid: 304 subjects received at least one dose of cadazolid and were included in the safety analysis. The median duration of treatment with cadazolid was 10 days.
- Vancomycin: 322 subjects received at least one dose of vancomycin and were included in the safety analysis. The median duration of treatment with vancomycin was 10 days.
Arm/Group | Cadazolid | Vancomycin
All-Cause Mortality (participants affected / at risk) | 7/304 | 7/322
Serious Adverse Events (participants affected / at risk) | 19/304 | 26/322
Other Adverse Events (participants affected / at risk) | 33/304 | 49/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cadazolid (N=304) | Vancomycin (N=322)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 8 (8)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rectal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cadazolid (N=304) | Vancomycin (N=322)
Abdominal pain (Gastrointestinal disorders) | 14 (16) | 22 (24)
Headache (Nervous system disorders) | 14 (17) | 25 (28)
Nausea (Gastrointestinal disorders) | 12 (13) | 24 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights.

DOCUMENTS (2):
  • Study Protocol (2015-10-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT01987895/Prot_001.pdf
  • Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT01987895/SAP_000.pdf